CLINICAL TRIAL: NCT06233630
Title: Erector Spinae Plane Block Vs. IPACK Block with Adductor Canal Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4/2024
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Anesthesia, Spinal; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Only spinal anaesthesia - No peripheral nerve block
  Interventions: Drug: Control Test - spinal anesthesia
- Erector Spinae Plane Block (Active Comparator): spinal anaesthesia and unilateral ultrasound guided erector spinae plane block - 20ml 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution ESPB
- Infiltration Popliteal Artery and Capsule of the Knee and Adductor Canal Block (Active Comparator): spinal anaesthesia and ultrasound guided Infiltration of local anesthetic between the Popliteal Artery and Capsule of the Knee (iPACK) block - 20ml 0.2% ropivacaine
  + ultrasound guided Adductor Canal Block - 10ml 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution iPACK+ACB

INTERVENTIONS:
Drug: Control Test - spinal anesthesia — No peripheral nerve block Only spinal anesthesia
  Other Names: spinal anesthesia
  Arms: Placebo
Drug: Ropivacaine 0.2% Injectable Solution ESPB — ultrasound guided erector spinae plane block (ESPB) - L2 level, unilateral
  Other Names: erector spinae plane block
  Arms: Erector Spinae Plane Block
Drug: Ropivacaine 0.2% Injectable Solution iPACK+ACB — ultrasound guided iPACK block + Adductor Canal Block
  Other Names: iPACK+ACB
  Arms: Infiltration Popliteal Artery and Capsule of the Knee and Adductor Canal Block

SUMMARY:
Effect of Erector Spinae Plane Block and iPACK block with Adductor Canal Block on pain management, and NLR and PLR following knee arthroplasty

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopedic procedures, especially in elderly patients, due to the deformation of joints. Patients may complain of severe pain due to surgical trauma and prosthesis. Regional anesthesia methods may be performed to reduce the inflammatory response, opioid consumption, and opioid-related side effects.

In recent years, the influence of regional anesthesiology on reducing the inflammatory response after surgical procedures has been emphasized. However, very few studies have evaluated the effect of various methods of anesthesia on the NLR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III,
* Aged 20-100 years,
* scheduled for knee arthroplasty under spinal anaesthesia

Exclusion Criteria:

* Patients who have a history of bleeding diathesis,
* Take anticoagulant therapy,
* have a History of chronic pain before surgery,
* have Multiple trauma,
* cannot assess their pain (dementia),
* have been operated on under general anaesthesia,
* have an infection in the area
* do not accept the procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 48 hours
  Total opiate consumption after surgery

SECONDARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 16 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 20 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
NLR | 24 hours postoperatively
  Neutrophil-to-lymphocyte ratio
PLR | 24 hours postoperatively
  Platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the medical research council muscle strength rating

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Domagalska, Ph.D., Principal Investigator — Poznan University of Medical Science
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No